CLINICAL TRIAL: NCT02023814
Title: Peripheral Blood CD34+ Cells Count as Predictor of Stem Cell Harvest After Chemotherapy and G-CSF. A Single Center Experience
Brief Title: Peripheral Blood CD34-positive Cells Enumeration as Predictor of Stem Cell Harvest
Status: Completed | Type: Observational
Sponsor: Ospedale Santa Croce-Carle Cuneo (Other)
Responsible Party: Principal Investigator, Roberto Sorasio, MD, Ospedale Santa Croce-Carle Cuneo
Other Study IDs: Emato_aferesi
Record Dates: First submitted 2013-12-19; First posted 2013-12-30 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-12

CONDITIONS: Blood Stem Cell Harvest Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study group: All patients who underwent stem cell mobilization after chemotherapy and G-CSF at our institution between 2002 and 2013

SUMMARY:
Stem cell mobilization procedures after chemotherapy and G-CSf performed at our Institution between 2002 and 2013 were reviewed in order to define prognostic factors for optimal harvest

ELIGIBILITY:
Inclusion Criteria:

* Mobilization with chemotherapy and G-CSF
* Years 2002-2013

Exclusion Criteria:

* mobilization with G-CSF alone
* mobilization with plerixafor

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent mobilization
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2002-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Blood Stem cell harvest failure rate | 7 days from hematological recovery
  Patients not able to harvest at least 2x10e6 CD34+/Kg in the specified time frame are considered failures

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Sorasio, Principal Investigator — Ospedale S Croce e Carle